CLINICAL TRIAL: NCT05728580
Title: Risk Factor for Percutaneous Coronary Intervention in the Beijing Friendship Hospital
Brief Title: PCI in Beijing Friendship Hospital
Acronym: BF-PCI
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BF-PCI
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-12

CONDITIONS: Cardiovascular Diseases; Percutaneous Coronary Intervention
Keywords: coronary heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to discover the potential risk factors related percutaneous coronary intervention. It aims to stratify the risk of PCI patients and discover the prognostic value of these risk fators.

DETAILED DESCRIPTION:
Coronary heart disease is the main cause of death worldwide. Ischemic heart disease is the most common cause of death. Percutaneous coronary intervention (PCI) is a very effective treatment for coronary heart disease, which can alleviate myocardial ischemia and reduce the mortality of patients with acute myocardial infarction. It is an important measure to treat coronary heart disease at present. However, the study found that the incidence of major adverse cardiac and cerebrovascular event (MACCE) after PCI was more than 10%, which could reach 20-30% in elderly patients. Therefore, the purpose of this study is to investigate the risk factors related to PCI and to intervene or change the treatment strategy as early as possible. Risk stratification was performed in these patients for improving the quality of life of patients, reducing medical costs, and improving the life expectancy of patients. Patients with PCI in Beijing friendship hospital are enrolled.The primary outcome is MACCE and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at the time of admission to the hospital
* PCI patients with coronary heart disease: according to the criteria interpreted in the 2011 American Guidelines for Percutaneous Coronary Intervention. The successful diagnostic criteria of PCI: residual stenosis of the treated vessel<10% (preferably 0%), and the forward flow is TIMI grade 3, there is no dissection that affects the flow, no important side branch occlusion, no visible thrombus and peripheral embolism.

Exclusion Criteria:

* Patients who failed in PCI treatment;
* Current known inability to follow instructions or comply with follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PCI accorrding to Inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-12-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
MACCE | These data is collected during follow-up for 5 years after discharge
  defined as a composite of all cause mortality, any myocardial infarction (MI), any revascularization, stroke, and heart failure hospitalization
All-cause mortality | These data is collected during follow-up for 5 years after discharge
  whether recidivation happened,whether other related disease happened

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Li, Dr, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided